CLINICAL TRIAL: NCT03603951
Title: A Phase 1 Study to Characterize Safety, Tolerance, Pharmacokinetics and Efficacy of SHR2554 in Subjects With Relapsed or Refractory Mature Lymphoid Neoplasms
Brief Title: A Phase 1 Study of SHR2554 in Subjects With Relapsed or Refractory Mature Lymphoid Neoplasms
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Collaborators: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR2554-I-101
Record Dates: First submitted 2018-07-10; First posted 2018-07-27 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Relapsed or Refractory Mature Lymphoid Neoplasms
Keywords: SHR2554; EZH2 inhibitor; phase 1; mature lymphoid neoplasm
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR2554 treated group (Experimental): Part I：treated with escalated doses of EZH2 inhibitor SHR2554 respectively； Part II：treated with fixed dose (RP2D) SHR2554 respectively
  Interventions: Drug: SHR2554

INTERVENTIONS:
Drug: SHR2554 — SHR2554 is a selective small molecule inhibitor of the histone-lysine methyltransferase EZH2.
  Other Names: EZH2 Inhibitor

SUMMARY:
This is a Phase 1 multicenter, single-arm, open-label, dose escalation and dose expansion study of enhancer of zeste homolog 2 (EZH2 ) inhibitor SHR2554.

This study will assess the tolerability, safety, pharmacokinetics, and preliminary anti-tumor activity of SHR2554 in participants with relapsed or refractory mature lymphoid neoplasms in part I, and the the efficacy in PTCL patients will be studied in Part II.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 70 years old (Adult, Senior)
2. Part I: Histologically or cytologically confirmed Mature lymphoid neoplasms; Part II: peripheral T cell lymphomas
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1；
4. Has a life expectancy of ≥12 weeks；
5. Resistant to standard therapy or no standard therapy available，have indications for treatment；
6. Have measurable disease （lymphoma participants，any nodes/nodal masses>1.5 cm in longest diameter (LDi) or extralymphatic sites of disease >1.0 cm in LDi；Multiple myeloma (MM) or Waldenström macroglobulinemia (WM) participants，serum M protein ≥0.5 g/dL or Bence Jones protein≥0.2 g/24 h）. （dose expansion study must satisfy）
7. Has sufficient tumor tissue (slides or blocks) available for testing EZH2 mutation status and expression level. （dose expansion study must satisfy）
8. Diffuse large B-cell lymphoma (DLBCL) participants have immunohistochemistry test results of cell origin (germinal center B-cell-like (GCB) or non-GCB), as well as myelocytomatosis oncogene (MYC), B cell lymphoma/leukemia 2 (BCL2) and B-cell lymphoma 6 (BCL6), or provide sufficient tumor tissue for testing. （dose expansion study must satisfy）
9. With adequate bone marrow function;
10. With adequate renal and liver function;
11. Coagulation function index：PT ≤1.5×ULN，APTT ≤1.5×ULN；
12. Women of childbearing potential (WOCBP) should be proven to be negative by human chorionic gonadotropin (hCG) test in 7 days before the first dose of SHR2554. They must be willing and able to employ a highly effective method of birth control/contraception to prevent pregnancy from the day they sign the informed consent form (ICF) to at least 30 days after receiving the last dose of study treatment. Male subjects with WOCBP partner should receive Surgical sterilization or consent to employ a highly effective method of birth control/contraception to prevent pregnancy；
13. Any prior treatment-related clinically significant toxicities have resolved to ≤ Grade 1 per CTCAE version 4.03 or prior treatment-related toxicities evaluated by physicians are not clinically significant at time of enrollment.
14. Participant who has provided written consent to participate in the study and ability to comply with all aspects of the protocol.

Exclusion Criteria:

1. Prior exposure to other inhibitor(s) of EZH2.
2. FL 3b or (potentially) transformed FL
3. Participants with a presence of central nerves invasion
4. Auto-transplantation within 60 days or allo-transplantation within 90 days before the first dose of study drug； >1 grade graft-versus-host disease (GVHD) or using GVHD control medicines that are not allowed by this trial；
5. Major surgery or serious trauma within 4 weeks before the first dose of study drug.；
6. anti-tumor agents within 4 weeks before the first dose of study drug（such as chemotherapy, radiotherapy, immunotherapy, target therapy and other clinical research）；Use of Chinese Herbal within 2 weeks before the first dose of study drug；use of Glucocorticoids to anti tumor within 7 days before the first dose of study drug（equivalent to prednisone>20 mg/d）；
7. Has known active infection with hepatitis B virus or hepatitis C virus（HBV DNA≥2×10^3 IU/mL，HCV RNA≥10^3 IU/mL）and liver dysfunction，need the intervention of anti-virus therapy;
8. Immunocompromised (i.e. has congenital immunodeficiency), including subjects known history of infection with human immunodeficiency virus (HIV) or has known active infection with tubercle bacillus；
9. Has an active infection or has a temperature > 38.5°C with unknown reasons（Investigators will decide the enrollment of participants with a fever that contributed to tumors）；
10. Has cardiovascular impairment，including history of congestive heart failure greater than New York Heart Association (NYHA) Class II, unstable angina, myocardial infarction, or stroke within 1 year prior to the planned first dose of study drug; or ventricular cardiac arrhythmia requiring medical treatment；
11. abnormal of ECG with clinical significance：such as prolongation of corrected QT interval using Fridericia's formula (QTcF)(male > 450 ms、female> 470 ms）；
12. History of cerebrovascular accident or transient ischemic attack within 6 months；
13. Has a prior malignancy other than the malignancies under study within 2 years- EXCEPTION: A subject with a history of a completely resected skin basal cell carcinoma, skin squamous-celled carcinoma, in situ cervical cancer or other in situ carcinomas, and has been relapse-free for 5 years；
14. Has serious acute/chronic disease or psychic disease，such as suicide intention or action in resent 1 year; or there are abnormal conditions that will increase the risk of using or managing study drug or affect the assessment of study results or investigator's judgment；
15. Staffs of institute sites directly related to the study or their family members, subordinates. Staffs of the sponsor pharmaceuticals company that directly related to the study；
16. Females who are pregnant or breastfeeding.
17. Inability to take oral medication, or any uncontrolled gastrointestinal condition (e.g., active gastroenteritis, chronic diarrhea, known diverticulosis, history of gastrectomy or gastric banding) that might impair the bioavailability of study drug. gastroesophageal reflux disease treated with proton pump inhibitors is eligible（should be no drug interaction）;
18. Use of known median or potent CYP3A4 or CYP3A5 inducers/inhibitors or P-gp inhibitors.
19. Any other major illness that, in the investigator's judgment, will substantially increase the risk associated with the subject's participation in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2018-08-14 (Actual); Primary Completion 2026-02-14 (Estimated); Study Completion 2026-08-14 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events (AEs) [Safety and Tolerability])（Part I） | through study completion, an average of about 6 months
  The incidence and severity of treatment-emergent AEs will be collected and the safety and tolerability of SHR2554 will be assessed.
Recommended phase 2 dose (RP2D)（Part I） | 30 days since the date of first dose
  Recommended phase 2 dose (RP2D) and/or maximum tolerated dose (MTD) will be established according to the incidence of dose-limiting toxicities (DLTs) of escalated doses of SHR2554.
Objective response rate (ORR)（Part II） | 60 days since the date of first dose
  assessed by independent radiology review committee (IRC)

SECONDARY OUTCOMES:
Time to peak (Tmax) | Day 1 and Day 2 of the single dose
  Pharmacokinetics profile of a single dose SHR2554 and its metabolite (plasma): Time to peak (Tmax) of plasma concentration
Maximum plasma concentration (Cmax) | Day 1 and Day 2 of the single dose
  Pharmacokinetics profile of a single dose SHR2554 and its metabolite (plasma): Maximum plasma concentration (Cmax)
Halflife (T1/2) | Day 1 and Day 2 of the single dose
  Pharmacokinetics profile of a single dose SHR2554 and its metabolite (plasma): Halflife (T1/2)
Clearance/ bioavailability (CL/F) | Day 1 and Day 2 of the single dose
  Pharmacokinetics profile of a single dose SHR2554 and its metabolite (plasma): Clearance/ bioavailability (CL/F)
apparent volume of distribution/bioavailability (Vd/F) | Day 1 and Day 2 of the single dose
  Pharmacokinetics profile of a single dose SHR2554 and its metabolite (plasma): apparent volume of distribution/bioavailability (Vd/F)
Area under curve (AUC) | Day 1 and Day 2 of the single dose
  Pharmacokinetics profile of a single dose SHR2554 and its metabolite (plasma): Area under curve (AUC)
Area under curve, steady state (AUCss) | Day 1 of cycle 1 to day 1 of cycle 4 (28 days/cycle)
  Pharmacokinetics profile of continuous medication of SHR2554 and its metabolite (plasma): Area under curve, steady state (AUCss)
Maximum plasma concentration, steady state (Cmax,ss) | Day 1 of cycle 1 to day 1 of cycle 4 (28 days/cycle)
  Pharmacokinetics profile of continuous medication of SHR2554 and its metabolite (plasma): Maximum plasma concentration, steady state (Cmax,ss)
Time to peak, steady state (Tmax,ss) | Day 1 of cycle 1 to day 1 of cycle 4 (28 days/cycle)
  Pharmacokinetics profile of continuous medication of SHR2554 and its metabolite (plasma): Time to peak, steady state (Tmax,ss)
Halflife (T1/2) | Day 1 of cycle 1 to day 1 of cycle 4 (28 days/cycle)
  Pharmacokinetics profile of continuous medication of SHR2554 and its metabolite (plasma): Halflife (T1/2)
Apparent volume of distribution, steady state/bioavailability (Vss/F) | Day 1 of cycle 1 to day 1 of cycle 4 (28 days/cycle)
  Pharmacokinetics profile of continuous medication of SHR2554 and its metabolite (plasma): Apparent volume of distribution, steady state/bioavailability (Vss/F)
Clearance/ bioavailability (CL/F) | Day 1 of cycle 1 to day 1 of cycle 4 (28 days/cycle)
  Pharmacokinetics profile of continuous medication of SHR2554 and its metabolite (plasma): Clearance/ bioavailability (CL/F)
Accumulation index (Rac) | Day 1 of cycle 1 to day 1 of cycle 4 (28 days/cycle)
  Pharmacokinetics profile of continuous medication of SHR2554 and its metabolite (plasma): Accumulation index (Rac)
Objective response rate (ORR) | every 8 weeks through study completion, an average of about 6 months
  Assess the response rate of subjects to the treatment of SHR2554
Progression-free survival (PFS) | every 8 weeks through study completion, an average of about 6 months
  Assess the survival condition of the subjects after the treatment of SHR2554
Duration of Response (DoR) | every 8 weeks through study completion, an average of about 6 months
  Assess the duration of complete/partial response after the treatment of SHR2554
Time to response（TTR）（Part II only） | 60 days since the date of first dose
  Assess the time to initial response of subjects to the treatment of SHR2554
OS（overall survival）（Part II only） | 2 years since the date of first dose
  Assess the overall survival of subjects treated by SHR2554

OTHER OUTCOMES:
Effect of escalated doses of SHR2554 on the histone H3 lysine 27 trimethylation (H3K27me3) level（Part I-exploratory endpoints） | day 1 of the single dose to day 1 of continuous medication cycle 2
  Analyze the level of H3K27me3 in the peripheral blood mononuclear cells of the subjects before and after the treatment of escalated doses of SHR2554.
EZH2 gene mutation（Part I-exploratory endpoints） | within 2 weeks after the last dose
  Assess the known mutation of EZH2 gene in tumor cells or tissues, analyze the relationship between efficacy and EZH2 mutation
EZH2 expression level（Part I-exploratory endpoints） | within 2 weeks after the last dose
  Assess EZH2 expression level in tumor tissues, analyze the relationship between efficacy and EZH2 expression level

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Peking University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Song Y, Jin Z, Li ZM, Liu Y, Li L, He C, Su H, Zhou H, Li K, Hao S, Zuo X, Wu J, Li D, Wu M, Sun X, Qi J, Cai Z, Li Z, Li Y, Huang Y, Shen J, Xiao Z, Zhu J. Enhancer of Zeste Homolog 2 Inhibitor SHR2554 in Relapsed or Refractory Peripheral T-cell Lymphoma: Data from the First-in-Human Phase I Study. Clin Cancer Res. 2024 Apr 1;30(7):1248-1255. doi: 10.1158/1078-0432.CCR-23-2582. PMID 38190117
- [Derived] Song Y, Liu Y, Li ZM, Li L, Su H, Jin Z, Zuo X, Wu J, Zhou H, Li K, He C, Zhou J, Qi J, Hao S, Cai Z, Li Y, Wang W, Zhang X, Zou J, Zhu J. SHR2554, an EZH2 inhibitor, in relapsed or refractory mature lymphoid neoplasms: a first-in-human, dose-escalation, dose-expansion, and clinical expansion phase 1 trial. Lancet Haematol. 2022 Jul;9(7):e493-e503. doi: 10.1016/S2352-3026(22)00134-X. PMID 35772429